CLINICAL TRIAL: NCT04347239
Title: A Phase 2b/3, Randomized, Double Blind, Placebo Controlled, Adaptive Design Study to Evaluate the Efficacy and Safety of Leronlimab for Patients With Severe or Critical Coronavirus Disease 2019 (COVID-19)
Brief Title: Evaluate the Efficacy & Safety of Leronlimab in Patients With Severe or Critical COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD12_COVID-19
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — leronlimab

STUDY DESIGN:
Intervention Model Description: There were 394 participants randomized to the blinded portion of the study using an Interactive Response Technology (IRT) system. A separate cohort of 90 new participants were enrolled in the open label portion of the study after completion of enrollment of the blinded portion.
  None of the participants involved in the blinded portion of the study were included in the open label portion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded pharmacists at clinical sites were notified of the arm to which the subjects were enrolled for the randomized portion of the study in order to prepare the appropriate treatment.
  There was no masking for the open-label portion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Syringes containing normal saline for injection were prepared by an unblinded pharmacist at the clinical sites for use as the placebo.
  Interventions: Drug: Placebo
- 700mg Leronlimab (Experimental): Each vial of active contains 350mg of leronlimab at a concentration of 175mg/ml (nominal 2mL fill volume) in formulation buffer containing histidine, glycine, sodium chloride, sorbitol, polysorbate 20 and sterile water for injections.
  Interventions: Drug: Leronlimab (700mg)
- 700mg Leronlimab Open Label (Experimental): Each vial of active contains 350mg of leronlimab at a concentration of 175mg/ml (nominal 2mL fill volume) in formulation buffer containing histidine, glycine, sodium chloride, sorbitol, polysorbate 20 and sterile water for injections.
  Interventions: Drug: Leronlimab (700mg)

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Leronlimab (700mg) — Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Other Names: PRO 140
  Arms: 700mg Leronlimab; 700mg Leronlimab Open Label

SUMMARY:
The purpose of this study was assess the safety and efficacy of leronlimab (PRO 140) administered as weekly subcutaneous injection in subjects with severe or critical COVID-19 disease.

DETAILED DESCRIPTION:
This was a Phase 2b/3, two-arm, randomized, double blind, placebo controlled, adaptive design multicenter study to evaluate the safety and efficacy of leronlimab (PRO 140) in patients with severe or critical symptoms of respiratory illness caused by coronavirus 2019 infection. Patients will be randomized to receive weekly doses of 700 mg leronlimab (PRO 140), or placebo. Leronlimab (PRO 140) and placebo will be administered via subcutaneous injection.

A single arm, non-randomized, open-label phase was added to the protocol after completion of enrollment in the randomized phase of the study.

The study had three phases: Screening Period, Treatment Period, and Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age at time of screening.
2. Subjects hospitalized with severe or critical illness caused by coronavirus 2019 infection as defined below:

   A. Severe Illness:

   - Diagnosed with COVID-19 by standard reverse transcriptase polymerase chain reaction (RT-PCR) assay or equivalent testing within 5 days of screening

   AND

   Symptoms of severe systemic illness/infection with COVID-19:

   - At least 1 of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath at rest or with exertion, confusion, or symptoms of severe lower respiratory symptoms including dyspnea at rest or respiratory distress

   AND

   Clinical signs indicative of severe systemic illness/infection with COVID-19, with at least 1 of the following:

   - respiration rate (RR) ≥ 30, heart rate (HR) ≥ 125, saturated oxygen (SaO2) <93% on room air or requires > 2L oxygen by nasal canula (NC) in order maintain SaO2 ≥93%, PaO2/FiO2 <300 (ratio of partial pressure of oxygen in arterial blood to fraction of inspired oxygen)

   AND

   - None of the following: Respiratory failure (defined by endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula, noninvasive positive pressure ventilation, or clinical diagnosis of respiratory failure in setting of resource limitations), Septic shock (defined by systolic blood pressure (SBP) < 90 mm Hg, or Diastolic BP < 60 mm Hg), Multiple organ dysfunction/failure

   B. Critical Illness:

   - Diagnosed with COVID-19 by standard RT-PCR assay or equivalent testing within 5 days of screening

   AND

   Evidence of critical illness, defined by at least 1 of the following:

   - Respiratory failure defined based on resource utilization requiring at least 1 of the following: Endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula, noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO), or clinical diagnosis of respiratory failure (in setting of resource limitation)

   OR

   - Shock (defined by SBP < 90 mm Hg, or Diastolic BP < 60 mm Hg or requiring vasopressors)

   OR

   -Multiple organ dysfunction/failure
3. Subject, if intubated, positive end expiratory pressure (PEEP) <15 cmH2O with PaO2/FiO2 >150 mmHg.
4. Electrocardiogram (ECG) with no clinically significant findings as assessed by the Investigator
5. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
6. Understands and agrees to comply with planned study procedures.
7. Women of childbearing potential and their partner must agree to use at least one highly effective method of contraception (e.g., hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], intrauterine devices, bilateral tubal occlusion, or sexual abstinence) for the duration of the study.

Exclusion Criteria:

1. Subjects with do-not-resuscitate (DNR) and/or do-not-intubate (DNI) orders or expected to be made DNR/DNI in setting of resource limitations or family wishes.
2. Not a candidate for dialysis or continuation of care (or full medical support) in setting of resource limitations.
3. Subject on continuous vasopressors (at the dose of norepinephrine >20μg/min and/or vasopressin >0.04 units/kg/min) for >48 hours at time of screening.
4. Subjects who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible.
5. Inability to provide informed consent or to comply with test requirements
6. Consideration by the investigator, for safety reasons, that the subject is an unsuitable candidate to receive study treatment
7. Pregnancy or breast feeding
8. Subject participating in another study with for an investigational treatment for COVID-19.

Note: Subject who were prescribed (1) hydroxychloroquine or chloroquine with or without azithromycin, (2) Remdesivir, (3) convalescent plasma therapy, or (4) immunomodulatory treatments (including but not limited to sarilumab, clazakizumab, tocilizumab, and anakinra) for the off-label treatment of COVID-19 prior to study enrollment may be included and may continue to receive these agents as part of standard-of-care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Study Director — CytoDyn, Inc.
Locations (18):
- United States (18):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - St. Jude Medical Center, Fullerton, California
  - UCLA, Los Angeles, California
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - Center for Advanced Research & Education (CARE), Gainesville, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Barnabas, Livingston, New Jersey
  - Atlantic Health System Hospital, Morristown, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Community Hospital of Brooklyn, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health, Winston-Salem, North Carolina
  - Ohio Health, Columbus, Ohio
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welch J, Dean J, Hartin J. Using NEWS2: an essential component of reliable clinical assessment. Clin Med (Lond). 2022 Nov;22(6):509-513. doi: 10.7861/clinmed.2022-0435. PMID 36427875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. First patient was enrolled into Part 1 of the study (blinded portion) on 16-April-2020. Data submitted represent analysis performed on data collected after all patients completed the Follow Up period.
Groups:
- Placebo: Two syringes each containing 2mL of normal saline for injection were prepared by an unblinded pharmacist at the clinical sites for use as the placebo.
- 700mg Leronlimab: Two syringes, each containing 350mg of leronlimab in 2mL, allowed administration of the 700mg dose, subcutaneously.
  Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
- 700mg Open Label: Two syringes each containing 350mg leronlimab
Period: Blinded Portion
Arm/Group | Placebo | 700mg Leronlimab | 700mg Open Label
Started | 129 | 265 | 0
Completed | 125 | 259 | 0
Not Completed | 4 | 6 | 0
Not completed — Pt randomized to study but withdrew consent before treatment with investigational product | 6 | 0 | 4
Period: Open Label
Arm/Group | Placebo | 700mg Leronlimab | 700mg Open Label
Started (Participants in the open-label portion of the study were only enrolled to the open label arm) | 0 | 0 | 90
Completed | 0 | 0 | 89
Not Completed | 0 | 0 | 1
Not completed — Pt enrolled but withdrew consent prior to dosing | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population is modified intent to treat population
Groups:
- 700mg Leronlimab - open label: Two syringes, each containing 350mg of leronlimab in 2mL, allowed administration of the 700mg dose, subcutaneously.
- Total: Total of all reporting groups
Arm/Group | 700mg Leronlimab | Placebo | 700mg Leronlimab - open label | Total
Number analyzed (Participants) | 259 | 125 | 89 | 473
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 171 | 96 | 57 | 324
  >=65 years | 88 | 29 | 32 | 149
Age, Continuous [Mean (Full Range); unit: years] | 58.82 [20 to 88] | 58.51 [28 to 86] | 59.18 [23 to 85] | 58.72 [20 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 42 | 25 | 157
  Male | 169 | 83 | 64 | 316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 11 | 7 | 1 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 29 | 23 | 17 | 69
  White | 133 | 70 | 54 | 257
  More than one race | 85 | 25 | 0 | 110
  Unknown or Not Reported | 0 | 0 | 17 | 17
Region of Enrollment [Number; unit: participants] — Study only enrolled patients in the US
  participants
    United States | 259 | 125 | 89 | 473
COVID SYMPTOM SCORE [Mean (Full Range); unit: units on a scale] — Ordinal scale assessment:
  1 = Death; 2 = Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4 = Hospitalized, requiring supplemental oxygen; 5 = Hospitalized, not requiring supplemental oxygen; 6 = Not hospitalized, limitation on activities; 7 = Not hospitalized, no limitations on activities.
  units on a scale | 3.2 [2.0 to 4.0] | 3.2 [2.0 to 4.0] | 3.3 [2.0 to 4.0] | 3.2 [2.0 to 4.0]

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality at Day 28
Description: Incidence of mortality at day 28
Time Frame: Mortality at day 28 (Visit 2, start of treatment = day 0)
Population: Modified Intent to Treat (mITT) population was used for the analysis. The mITT population is defined as the set of subjects who randomized and have received at least one dose of leronlimab (PRO 140) or placebo. This population was used for the primary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- 700mg Open Label: Two syringes, each containing 350mg leronlimab administered once weekly for 2 weeks.
Arm/Group | 700mg Leronlimab | Placebo | 700mg Open Label
Number analyzed (Participants) | 259 | 125 | 89
Participants
  Mortality | 52 | 27 | 23
  Survival | 207 | 98 | 66

2. Secondary Outcome: All-cause Mortality at Day 14
Description: Day 0 refers to the data of randomization/first treatment.
Time Frame: Mortality at day 14 (initiation of treatment = day 0)
Population: Modified Intent to Treat (mITT) population was used for the analysis. The mITT population is defined as the set of subjects who randomized and have received at least one dose of leronlimab (PRO 140) or placebo. This population was used for the secondary outcome endpoint analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 700mg open label: Two syringes each containing 350mg leronlimab, once weekly for two weeks
Arm/Group | 700mg Leronlimab | Placebo | 700mg open label
Number analyzed (Participants) | 259 | 125 | 89
Participants | 25 | 13 | 17

3. Secondary Outcome: Proportion of Patients Achieving a Category of 6 or Higher on the Ordinal Scale at Days 14 and 28 (on a 7 Point Ordinal Scale).
Description: Evaluation of the clinical status of participants at Day 28 was assessed with a 7-level ordinal scale (OS) (with higher score indicating better outcome).
  The OS of patient health status ranged from: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. The study enrolled hospitalized patients with an OS Score of 2, 3, or 4 at baseline. The OS score of 6 refers to a participant who is not hospitalized with limitation on activities and 7 refers to not hospitalized with no limitations on activities.
Time Frame: Change from baseline to days 14 and 28
Population: Responders refer to subjects who achieved a category of 6 or higher at Day 14 and/or Day 28. Note: Proportions are based on the result of multiple imputation.
Measure: Number; unit: Proportion of patients
Groups:
- Placebo: Syringes containing normal saline for injection were prepared by an unblinded pharmacist at the clinical sites for use as the placebo.
  Placebos: Placebo
Arm/Group | 700mg Leronlimab | Placebo | 700mg Open Label
Number analyzed (Participants) | 259 | 125 | 89
Proportion of patients
  Responders at d28 | 0.58 | 0.55 | 0.46
  Non-responders at d28 | 0.41 | 0.45 | 0.47
  Missing at d28 | 0 | 0 | 0.07
  Responders at d14 | 0.38 | 0.42 | 0.39
  Non-responders at d14 | 0.62 | 0.58 | 0.47
  Missing at D14 | 0 | 0 | 0.13

4. Secondary Outcome: Change in Clinical Status of Subjects at Day 28 (on a 7 Point Ordinal Scale)
Description: Evaluation of the clinical status of participants at Day 28 was assessed with a 7-level ordinal scale (OS) (with higher score indicating better outcome).
  The OS of patient health status ranged from: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. The study enrolled hospitalized patients with an OS Score of 2, 3, or 4 at baseline.
  Baseline is last available value before treatment. Change from baseline is based on patients with paired values. The p value is from rank ANCOVA model adjusted for stratification factor and age using imputed data. All results and change from baseline are based on the result of multiple imputation.
Time Frame: Change from start of treatment (baseline) to day 28
Population: Rank ANCOVA model adjusted for stratification factor and age based on non-missing observed data. Change from baseline is based on patients with paired values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 700mg Leronlimab | Placebo | 700mg Open Label
Number analyzed (Participants) | 259 | 125 | 89
score on a scale | 1.5 (2.25) | 1.4 (2.18) | 1.0 (2.1)

5. Secondary Outcome: Length of Hospital Stay
Description: Length of Hospital Stay measured in days
Time Frame: Timeframe is from screening visit to end of treatment (visit 5)
Population: Modified Intent to Treat (mITT) population was used for the analysis. The mITT population is defined as the set of subjects who randomized and have received at least one dose of leronlimab (PRO 140) or placebo. Patients with incomplete data were excluded from the analysis. This population was used for the secondary outcome endpoint analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | 700mg Leronlimab | Placebo | 700mg Open Label
Number analyzed (Participants) | 259 | 125 | 74
Days | 15 [1 to 45] | 14 [1 to 46] | 14 [1 to 45]

6. Other Pre Specified Outcome: All-Cause Mortality at Day 14 in the Critically Ill Population
Description: All-cause mortality at day 14 in the critically ill population. Day 0 refers to the date of randomization/first treatment.
Time Frame: Mortality at day 14 (initiation of treatment = day 0)
Population: There were 62 patients in the critically ill population. Critically ill was defined as patients that were hospitalized, on invasive ventilation or extracorporeal membrane oxygenation (ECMO). Critically ill subjects were a subgroup of the Modified Intent to Treat population used for this analysis. As defined in the SAP, subgroup analysis was performed on predefined stratification factors including the subgroup of patients identified as "critically ill" and defined as above.
Measure: Count of Participants; unit: Participants
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 43 | 19
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Study drug was administered at Visit 2 (day 0) and visit 4 (day 7). Adverse events and medications were monitored throughout the study from Visit 2 (day 0, first treatment) through completion of follow up which is Visit 7, (4 weeks after the End of Treatment visit) for a total of 42 days.
Arm/Group | Placebo | 700mg Leronlimab | 700mg Open Label
All-Cause Mortality (participants affected / at risk) | 31/125 | 60/259 | 23/89
Serious Adverse Events (participants affected / at risk) | 47/125 | 99/259 | 35/89
Other Adverse Events (participants affected / at risk) | 77/125 | 142/259 | 29/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | 700mg Leronlimab (N=259) | 700mg Open Label (N=89)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 23 (26) | 61 (73) | 30 (40)
Infections and Infestations (Infections and infestations) | 25 (27) | 38 (39) | 10 (13)
Cardiac Disorders (Cardiac disorders) | 12 (12) | 22 (26) | 7 (10)
Renal and Urinary Disorders (Renal and urinary disorders) | 12 (12) | 16 (16) | 4 (4)
Investigations (Investigations) | 3 (3) | 7 (8) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 4 (4) | 6 (7) | 1 (1)
Metabolism and Nutrition (Metabolism and nutrition disorders) | 3 (4) | 6 (6) | 2 (3)
Gen Disorders and Admin Site Conditions (General disorders) | 3 (3) | 5 (5) | 0 (0)
Blood and Lymph (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0)
Hepatobiliary (Hepatobiliary disorders) | 1 (1) | 3 (4) | 0 (0)
Vascular Disorders (Vascular disorders) | 0 (0) | 4 (4) | 3 (4)
Musculoskeletal and Connective Tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | 700mg Leronlimab (N=259) | 700mg Open Label (N=89)
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 33 (46) | 76 (104) | 13 (18)
Infections And Infestations (Infections and infestations) | 34 (53) | 60 (85) | 12 (20)
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 21 (32) | 46 (76) | 12 (18)
Cardiac Disorders (Cardiac disorders) | 21 (25) | 36 (50) | 10 (14)
Investigations (Investigations) | 23 (28) | 26 (43) | 1 (1)
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 15 (19) | 27 (41) | 5 (10)
Vascular Disorders (Vascular disorders) | 17 (25) | 21 (26) | 5 (9)
Renal And Urinary Disorders (Renal and urinary disorders) | 15 (17) | 30 (31) | 5 (6)
Gastrointestinal Disorders (Gastrointestinal disorders) | 18 (26) | 17 (22) | 4 (4)
Nervous System Disorders (Nervous system disorders) | 14 (17) | 15 (22) | 2 (5)
General Disorders And Administration Site Conditions (General disorders) | 14 (16) | 12 (14) | 4 (4)

LIMITATIONS AND CAVEATS:
The outcome and safety data came from a report from the contract research organization that oversaw the study. A review of 64 Case Report Forms for the open label portion of the study indicated that over 70% contained no information about adverse events, therefore the adverse events for the open label portion of the study may be underreported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT04347239/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04347239/SAP_001.pdf
  • Informed Consent Form (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT04347239/ICF_002.pdf